CLINICAL TRIAL: NCT04710472
Title: Randomized Controlled Trial of a Mobile App for Remote Patient Monitoring in Oncology: a Phase II Trial
Brief Title: MentorApp for Cancer Patient's Remote Monitoring
Acronym: MentorA1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associacao de Investigacao de Cuidados de Suporte em Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AICSO3
Record Dates: First submitted 2021-01-10; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: cancer; supportive care; digital healthcare; remote monitoring; symptoms; quality of life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MH (Experimental): Arm MH - mobile Mentora app to monitor and track treatment side-effects, vital signs, therapeutics and daily habits;
  Interventions: Device: Mentora App
- C (No Intervention): SOC

INTERVENTIONS:
Device: Mentora App — Participants will be invited to register their treatment side effects, symptoms, daily activities and exercise and QoL on a health app designed for this purpose.
  The Mentora Health App includes a tool based on PRO-CTCAE™, a patient-reported outcome measurement system developed by the National Cancer Institute, version 1.1, that includes 80 symptoms (attachment 1) and has been translated and validated to Portuguese (Portugal) by the authoring entity. These symptoms are graded on a five-point scale from 0 (not present) to 4 (disabling) based on clinical criteria.
  Arms: MH

SUMMARY:
With the growing number of cancer survivors, challenges to deal with comorbidities and impacted quality of life of cancer survivors by the disease and treatments also surge. Symptoms and Adverse Events are common and insufficiently monitored in real time / real life, which leads to increased symptom burden, treatment delays and unplanned hospital admissions. Remote monitoring apps have been shown to improve quality of life, symptom control and survival in published clinical trials, but no data with such interventions exists on the Portuguese population.

A phase II randomized controlled trial to explore the feasibility of a mobile app for remote symptom monitoring in cancer patients will be done. Patients will be recruited in Portuguese Hospitals and will be invited to test the app for three months. Patient experience and satisfaction will be assessed via a weekly survey. Quality of life will be assessed at 1 and 3 months.

The results of this pilot study will inform subsequent randomized clinical trials to test safety and efficacy of remote monitoring and lifestyle interventions to improve symptoms control and quality of life.

DETAILED DESCRIPTION:
The primary aim is to assess the feasibility and usability of a mobile app (MHapp) to remote register and monitor treatment side effects, lifestyle habits and clinical data in cancer patients.

This is a phase II randomized controlled trial with two study arms:

Arm MH - mobile Mentora app to monitor and track treatment side-effects, vital signs, therapeutics and daily habits; Arm C - SOC

No sham intervention is thought to be viable as we want to test the MHapp as a whole complex intervention with all different components and compare it with current SOC. Patients will be screened at oncology visits for inclusion criteria. It is not viable also to blind clinicians once the app provides a detailed progress report of which we want to assess the impact on oncology care and clinical team satisfaction. We will blind statisticians and people performing the final analysis.

Once agreeing to enrol, patients will be randomly allocated to one of the study arms through a computer generated sequence of numbers, concealed from the clinical staff and patients.

8.1 Study design and Population

Randomized controlled clinical trial with two arms - arm MH (intervention with the MH app) and arm C (controls - standard of care). We will recruit 50 cancer patients in systemic treatments in Portuguese hospitals with oncology service.

Inclusion criteria:

adults (18 years old or older) with a cancer diagnosis at any stage Receiving systemic chemotherapy not in the context of a clinical trial, with treatment expected to continue for at least three months counting from time of enrollment fluent in written Portuguese with a personal mobile smartphone (android or iphone any version) willing to give informed consent for study participation

Exclusion criteria:

Cognitive impairment or disability that limits capacity to comply with study interventions and assessments Having a life expectancy < 3 months as determined by the attending oncologist ECOG performance status greater than 2 Unable to read and comprehend portuguese language text Participants will remain on study until discontinuation of cancer treatment, voluntary withdrawal, or death.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 years old or older)
* with a cancer diagnosis at any stage
* Receiving systemic chemotherapy not in the context of a clinical trial, with treatment
* expected to continue for at least three months counting from time of enrollment
* fluent in written Portuguese
* with a personal mobile smartphone (android or iphone any version)
* willing to give informed consent for study participation

Exclusion Criteria:

* Cognitive impairment or disability that limits capacity to comply with study interventions and assessments
* Having a life expectancy < 3 months as determined by the attending oncologist
* ECOG performance status greater than 2
* Unable to read and comprehend portuguese language text

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
feasibility and usability of the MHapp | 1 month
  The outcome will be considered positive if at least one of the 2 following criteria applies to more than 60 percent of participants enrolled:
  replies to 2 or more weekly reports OR at least one weekly log in to the app.

SECONDARY OUTCOMES:
To evaluate the impact of MHapp on cancer patients QoL on European Organisation for Research and Treatment of Cancer.(EORTC) Core (c)30 | 1 and 3 months
  Impact of MHapp on cancer Qol
To explore the satisfaction of cancer patients, clinical teams and their carers with the MHapp | 1 week, 1 month, 3 months
  Patient's satisfaction with the app will be documented via survey at 1 week, 1 month and 3 months from D1 and interview at 1 month; Satisfaction of clinical oncology doctors and nurses with the information report provided by the MHapp on a Likert scale from 0 (not satisfied at all) to 7 (Very satisfied) and through qualitative analysis of open ended questions via interview at the end of the study period
To understand how to improve users' experience navigating the MHapp | 1 week, 1 month, 3 months
  General question about usability and ease of use will be asked on the survey done at 1 week, 1 month and 3 months from D1 and explored in further detail at the interview at 1 month;
To report adherence rates to the app usage at 1 and 3 months on the intervention arm | 1 month, 3 months
  Percentage of side effects and adverse events reported on medical appointments also registered in the MHapp during the 1st month on study Total attendance - retention rate/total withdraw from study (30 days)
To compare healthcare resources use in both study arms | 1 month, 3 months
  Report healthcare resources use:
  number of unplanned hospital visits or calls; unplanned hospitalizations; time inside medical appointments.
To evaluate the impact on AEs G>2 per CTCAE (Common Terminology Criteria for Adverse Events) v.5 (minimum 1 maximum 4) | 1 and 3 months
  Frequency of G>2 AEs

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Ribeiro, Principal Investigator — Associacao de Investigacao de Cuidados de Suporte em Oncologia